CLINICAL TRIAL: NCT03114852
Title: The REGENT Study: Familiar Renal Disease, Epidemiology and Genetics in Niteroi/Rio de Janeiro
Brief Title: Familiar Renal Disease, Epidemiology and Genetics in Niteroi/Rio de Janeiro
Acronym: REGENT
Status: Completed | Type: Observational
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Jorge R Almeida, MD, Professor, Universidade Federal Fluminense
Other Study IDs: REGENT study
Record Dates: First submitted 2017-03-20; First posted 2017-04-14 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2019-08

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood collection of patients with familial history of renal disease will be done to extract DNA and to perform analysis of mutations and sequencing. After that, the samples will not be retained.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CKD patients: 'blood collection'
  Patients with chronic kidney disease in renal replacement therapy living in the sanitary administrative region of Niteroi/Rio de Janeiro. They will be interviewed about past history of familiar renal disease. They will have blood functional renal biochemistry analysed.
  Interventions: Diagnostic Test: blood collection
- Renal Familiar Disease: 'blood collection' They will have blood tested to renal genetic diseases
  Interventions: Diagnostic Test: blood collection

INTERVENTIONS:
Diagnostic Test: blood collection — They will have blood tested to renal genetic diseases

SUMMARY:
The REGENT study (Familiar Renal Disease, Epidemiology and Genetics in Niteroi/Rio de Janeiro) is a epidemiological study that try to identify and clinically describe questions about genetic renal diseases in a southeast Brazilian population undergoing renal replacement therapy.

DETAILED DESCRIPTION:
In Brazil, several kidney diseases have unknown etiological diagnosis, among them, hereditary renal diseases. The lack of technical-scientific knowledge and patients' access to the health service hinder the correct diagnosis, so that hundreds of patients with chronic kidney disease (CKD) are unaware of the origin of their kidney problems. The objective of this REGENT study (Renal epidemiology and genetics in Niteroi) is to identify and characterize the cases of possible inheritance of CKD in patients undergoing dialysis or kidney transplant treatment in the metropolitan region II of the state of Rio de Janeiro. In this metropolitan region, based in the city of Niteroi, there are 10 hemodialysis clinics accounting for approximately 1500 - 1800 patients. There is a central Hospital that works as an official reference center for all those CKD patients (Hospital Universitario Antonio Pedro). This hospital belongs to the Universidade Federal Fluminense, an academic research institution, where this project will be executed. There is also a kidney transplant unit working at the Hospital Universitario Antonio Pedro. Interviews, sociodemographic and clinical data collection will be performed in patients with CKD from these centers. The interview contains questions about family CKD: Does any family member undergo hemodialysis or peritoneal dialysis? Does any family member do/did conservative treatment for CKD? Has any family member had a kidney transplant? Has any family member died due to chronic kidney disease? In cases of any affirmative answer to one of the above questions, patients will be classified as a "family index case". The cases of familial kidney disease caused by diabetes, and polycystic kidney disease will be excluded. So, the remaining cases will be considered as "index cases" to be more described and characterized. In this way, an affirmative response to the survey will create a group of familial CKD, and it will allow us to identify them as a suspected genetic kidney disease. These patients will be analyzed as a group, and clinical histories and blood tests to genetic renal diseases will also be performed, when possible, depending on the availability. From these identified index cases, we will try to create familiar clinical description of each individual in every family. A new outpatient section is being created at the Hospital Universitario Antonio Pedro to take multidisciplinary care of the relatives and entire families in a special type of family primary care.

ELIGIBILITY:
Inclusion Criteria:

* Brazilian patients underwent any type of renal replacement therapy, dialysis or kidney transplantation living in the area of Niteroi/Rio de Janeiro.
* Relatives among the familial people of the index cases.

Exclusion Criteria:

* Diabetic Nephropathy
* Non-familial cases of known Glomerulonephritis
* Refuse in participating of interview and blood collection to genetic tests

Ages: 12 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population to be studied will be formed by southeast Brazilians that are on renal replacement therapy as dialysis or kidney transplantation. Such patients with renal diseases will answer a questionnaire about familial involvement. Some of them will be characterized as a familial index case of not yet determined genetic kidney disease.
Sampling Method: Non-Probability Sample
Enrollment: 1308 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-09-19 (Actual)

PRIMARY OUTCOMES:
Frequency and numbers of patients with renal familial diseases that are on renal replacement therapy in southeast Brazil. | The familial epidemiological results will be ready up to 24 months form the start of the study.
  We will proceed a clinical interview using a questionnaire focused on the family history, among each Brazilian patients from dialysis or transplant center from the region of Niteroi/Rio de Janeiro. Patients with a positive history of familial disease will be included as a "case of familial renal disease". The results of the interviews will be analysed to create a report about incidence and prevalence of genetic renal disease among the southeast Brazilian people. At the same time we are creating a genetic reservoir to characterization of renal diseases in southeast of Brazil and we are also creating the basis to a cohort study based these families, through a new recently created outpatient unit to take care of familial renal diseases to follow all these involved renal families.

SECONDARY OUTCOMES:
Frequency of uromodulin and APOL-1 mutation in southeast Brazilian patients underwent renal replacement therapy | From the time to DNA extraction, by using molecular studies, the DNA samples of each index cases will be analyised to uromodulin and APOL1, up to 48 months.
  A complete mutation analysis, with identification of polimorphism SNPs to uromodulin and APOL-1 will be place as an initial specific protocol by using extracted DNA from the familial index cases.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge R Almeida, MD, PhD, Principal Investigator — Universidade Federal Fluminense
Locations (1):
- Universidade Federal Fluminense, Niterói, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided